CLINICAL TRIAL: NCT03908632
Title: An Observational Study to Assess the Prevalence and Outcomes of Primary Pulmonary Coccidioidomycosis in Persons Aged > / = 14 Years Presenting With Community Acquired Pneumonia (CAP) in Endemic Areas (SAnds-PPC)
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-1053
Record Dates: First submitted 2019-03-27; First posted 2019-04-09 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2022-07-25

CONDITIONS: Coccidioidomycosis; Pneumonia
Keywords: Community Acquired Pneumonia; Endemic Areas; Observational Study; Primary Pulmonary Coccidioidomycosis
MeSH Terms: conditions — Coccidioidomycosis; Pneumonia; Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples (approximately 10 mL) to determine Coccidioides antibodies for entry will be performed locally at the sites for Step 1 Day 1, and if negative this will be repeated at Day 22. Erythrocyte sedimentation rate (ESR), high sensitivity C-reactive protein (hsCRP), and procalcitonin will be measured on Step 1 Day 1, or if enrolled directly into Step 2, at Step 2 Day 1. Total blood volume for subjects participating only in Step 1 will be up to 65 ml (95 mL for subjects consenting to additional sample collection for future use). Total blood volume collected per participant who participates in Step 1 and Step 2 is up to 95 mL (up to 155 mL for subjects consenting to additional sample collection for future use). Volumes may be higher for subjects with additional clinic visits after Step 2 Visit 06 due to persistent or disseminated disease.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Step 1: Subjects 14 years or older diagnosed with Community Acquired Pneumonia (CAP) and positive serology for primary pulmonary coccidioidomycosis (PPC) will enroll in Step 1 within 14 days of symptom onset, n=750
- Step 2: Subjects with a diagnosis of primary pulmonary coccidioidomycosis (PPC) confirmed by positive serologic testing during Step 1 will enter Step 2 within 21 days of their test collection date, n=200

SUMMARY:
This is an observational study in 750 individuals aged 14 years or older, diagnosed with Community Acquired Pneumonia (CAP) who meet all eligibility criteria in Coccidioides endemic regions. This study is designed to provide data on the prevalence of primary pulmonary coccidioidomycosis among persons presenting with CAP in endemic regions. Among individuals diagnosed with primary pulmonary coccidioidomycosis, we aim to describe the clinical course, predictors of the clinical course and compare the response to prescribed antifungal therapy versus no antifungal therapy. The hypothesis for patients with primary pulmonary coccidioidomycosis is that early treatment with antifungal therapy is effective in reducing the frequency, severity and associated adverse outcomes of infection with recently acquired coccidioidomycosis pneumonia. The study will be divided into Step 1 and Step 2. Step 1 will identify which subjects have primary pulmonary coccidioidomycosis based on the case definition for the protocol and Step 2 will follow subjects who meet the case definition and will observe their clinical management and clinical outcomes. Subjects will enroll in Step 1 within 28 days of symptom onset. In Step 1, blood work for serologic determination of Coccidioides infection will be drawn at the time of enrollment (Day 1), and again 21 days later if a positive result is not reported at Day 1. Subjects with a diagnosis of primary pulmonary coccidioidomycosis confirmed by positive serologic testing during Step 1 will enter Step 2 within 21 days of a positive test result; subjects with a negative serology at Day 1 and Day 22 will not be followed further. Subjects referred to the study after a diagnosis of primary pulmonary coccidioidomycosis confirmed by positive serologic testing will also be allowed to enter Step 2 directly within 21 days of a positive test result and within 7 weeks of symptom onset, as long as they meet study enrollment criteria. The primary objective is to assess the prevalence of primary pulmonary coccidioidomycosis (PPC) in subjects with community acquired pneumonia (CAP) in coccidioidomycosis endemic areas.

DETAILED DESCRIPTION:
This is an observational study in 750 individuals aged 14 years or older, diagnosed with Community Acquired Pneumonia (CAP) who meet all eligibility criteria in Coccidioides endemic regions. This study is designed to provide data on the prevalence of primary pulmonary coccidioidomycosis among persons presenting with CAP in endemic regions. Among individuals diagnosed with primary pulmonary coccidioidomycosis, we aim to describe the clinical course, predictors of the clinical course and compare the response to prescribed antifungal therapy versus no antifungal therapy. The hypothesis for patients with primary pulmonary coccidioidomycosis is that early treatment with antifungal therapy is effective in reducing the frequency, severity and associated adverse outcomes of infection with recently acquired coccidioidomycosis pneumonia. The study will be divided into Step 1 and Step 2. Step 1 will identify which subjects have primary pulmonary coccidioidomycosis based on the case definition for the protocol and Step 2 will follow subjects who meet the case definition and will observe their clinical management and clinical outcomes. Subjects will enroll in Step 1 within 28 days of symptom onset. In Step 1, blood work for serologic determination of Coccidioides infection will be drawn at the time of enrollment (Day 1), and again 21 days later if a positive result is not reported at Day 1. Subjects with a diagnosis of primary pulmonary coccidioidomycosis confirmed by positive serologic testing during Step 1 will enter Step 2 within 21 days of a positive test result; subjects with a negative serology at Day 1 and Day 22 will not be followed further. Subjects referred to the study after a diagnosis of primary pulmonary coccidioidomycosis confirmed by positive serologic testing will also be allowed to enter Step 2 directly within 21 days of a positive test result and within 7 weeks of symptom onset, as long as they meet study enrollment criteria. The primary objective is to assess the prevalence of primary pulmonary coccidioidomycosis (PPC) in subjects with community acquired pneumonia (CAP) in coccidioidomycosis endemic areas. The secondary objectives are divided into two categories. For subjects with CAP in coccidioidomycosis endemic areas the secondary objectives are: 1) To determine demographic, clinical and laboratory factors that predict PPC; 2) To describe the practice of empiric antifungal treatment of subjects with CAP. For subjects with confirmed primary pulmonary coccidioidomycosis the secondary objectives are: 1) To describe the clinical course of primary pulmonary coccidioidomycosis from earliest presentation; 2) To assess the demographic, clinical, laboratory and treatment predictors of the clinical course of primary pulmonary coccidioidomycosis; 3) To describe the practice of antifungal treatment of subjects with confirmed primary pulmonary coccidioidomycosis; 4) To compare the outcomes of antifungal therapy vs. no therapy for primary pulmonary coccidioidomycosis as measured by clinical signs and symptoms, functional scores of health and well-being and ability to participate in social roles and activities, time missed from school and work, dissemination, and mortality.

ELIGIBILITY:
Inclusion Criteria:

Step 1 Subject Inclusion Criteria:

1. Aged > / = 14 years and presenting for clinical care in coccidioidomycosis endemic areas.
2. Diagnosis of community acquired pneumonia (CAP) established by a health care provider.
3. Pulmonary opacity on chest X-ray or computerized tomography (CT) scan consistent with CAP.
4. Onset of symptoms related to current CAP diagnosis within 28 days prior to enrollment.
5. Must be able to understand the study and provide informed consent.*

   *If aged < 18 years, the parent(s) or guardian must be able to understand the study and provide informed consent, with the assent of the minor.
6. Willing and able to comply with study procedures and complete study visits.
7. Willing to allow access to medical records, and medical records are available to the study team.

Step 2 Subject Inclusion Criteria:

1. Aged > / = 14 years
2. Presence of at least one influenza-like sign or symptom (e.g. fever, chest pain, cough, myalgia, arthralgia, and headache.
3. Onset of any symptoms no earlier than 7 weeks prior to enrollment into Step 2.
4. Opacity/pleural effusion diagnosed by chest radiograph or computerized tomography (CT) scan .
5. Positive result for any serologic test confirming coccidioidomycosis obtained within 21 days prior to enrollment into Step 2.*

   * The assays considered for this criterion are: coccidioidal immunoglobulin M (IgM) by immunodiffusion, enzyme immunoassay (EIA), latex agglutination or tube precipitin OR coccidioidal immunoglobulin G (IgG) by immunodiffusion, EIA, or complement fixation. The interpretation of positive or negative is per the reporting laboratory instructions
6. Must be able to understand the study and provide informed consent.**

   **If aged <18 years, the parent(s) or guardian must be able to understand the study and provide informed consent, with the assent of the minor.
7. Willing and able to comply with study procedures and complete study visits.
8. Willing to allow access to medical records, and medical records are available to the study team.

Exclusion Criteria:

Step 1 Subject Exclusion Criteria:

1. Have documented microbiologically- or serologically-confirmed past infections with Coccidioides.*

   *An initial positive serologic test obtained within 21 days inclusive prior to enrollment is permissible.
2. Hospitalization within 14 days prior to the onset of pneumonia symptoms.
3. Presence of cavitary lung disease.
4. Evidence of disseminated, extrathoracic disease.

Step 2 Subject Exclusion Criteria:

1. Have documented microbiologically- or serologically-confirmed past infections with Coccidioides.*

   *An initial positive serologic test obtained within 21 days inclusive prior to enrollment is permissible.
2. Presence of cavitary lung disease.
3. Evidence of disseminated, extrathoracic disease.

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Step 1 will include at least 750 persons aged 14 and older diagnosed with community acquired pneumonia (CAP) in coccidioidomycosis endemic areas. Step 2 will involve at least 200 persons aged 14 and older with primary pulmonary coccidioidomycosis.
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-05 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with primary pulmonary coccidioidomycosis (PPC) among subjects with Community Acquired Pneumonia CAP) in Step 1 | Day 1 through Day 22

SECONDARY OUTCOMES:
Associations between chest radiograph and antifungal treatment for PPC, Step 2 | Day 1 through Day 730
Associations between Observational Study to Assess the Prevalence and Outcomes of Primary Pulmonary Coccidioidomycosis (SAnds-PPC) and antifungal treatment for PPC, Step 2 | Day 1 through Day 730
Associations between severity and antifungal treatment for PPC, Step 2 | Day 1 through Day 730
Compare change in chest radiograph findings score for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 1 through Day 730
Compare disease severity score for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 1 through Day 365
Compare mortality rates for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 1 through Day 365
Compare percent of subjects that develop persistent or disseminated PPC for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 85 through Day 730
Compare SAnds-PPC score for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 1 through Day 730
Compare time missed from school and work for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 1 through Day 180
Descriptive statistics of subjects' demographics in Step 1 | Day 1
Descriptive statistics of subjects' Erythrocyte Sedimentation Rate (ESR) in Step 1 | Day 1
Descriptive statistics of subjects' High sensitivity C-reactive protein (hsCRP) in Step 1 | Day 1
Descriptive statistics of subjects' Observational Study to Assess the Prevalence and Outcomes of Primary Pulmonary Coccidioidomycosis (SAnds-PPC) in Step 1 | Day 1
Descriptive statistics of subjects' procalcitonin in Step 1 | Day 1
Descriptive statistics of subjects' serologic titers in Step 1 | Day 1
Frequency of prescription of antifungal therapy prescribed for Community Acquired Pneumonia (CAP) for Step 1 | Day 1 through Day 22
Frequency of prescription of antifungal therapy prescribed for primary pulmonary coccidioidomycosis (PPC) for Step 2 | Day 1 through Day 730
Mean of change in chest radiograph findings score as a part of standard of care, Step 2 | From 4 to 8 weeks after Initial chest x-ray date
Mean of disease severity score for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Mean of the disease severity score for subjects with persistent or disseminated primary pulmonary coccidioidomycosis (PPC), Step 2 | Day 180 through Day 365
Mean of the modified SAnds-PPC score (clinical scoring system) for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Mean of the SAnds-PPC score (clinical scoring system) for subjects with persistent or disseminated primary pulmonary coccidioidomycosis (PPC), Step 2 | Day 180 through Day 365
Mean of time to resolution of each symptom contributing to the modified SAnds-PPC score for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Median of change in chest radiograph findings score as a part of standard of care, Step 2 | From 4 to 8 weeks after Initial chest x-ray date
Median of disease severity score for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Median of the disease severity score for subjects with persistent or disseminated primary pulmonary coccidioidomycosis (PPC), Step 2 | Day 180 through Day 365
Median of the modified SAnds-PPC score (clinical scoring system) for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Median of the SAnds-PPC score (clinical scoring system) for subjects with persistent or disseminated primary pulmonary coccidioidomycosis (PPC), Step 2 | Day 180 through Day 365
Median of time to resolution of each symptom contributing to the modified SAnds-PPC score for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Quartiles of change in chest radiograph findings score as a part of standard of care, Step 2 | From 4 to 8 weeks after Initial chest x-ray date
Quartiles of disease severity score for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Quartiles of the disease severity score for subjects with persistent or disseminated primary pulmonary coccidioidomycosis (PPC), Step 2 | Day 180 through Day 365
Quartiles of the modified SAnds-PPC score (clinical scoring system) for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Quartiles of the SAnds-PPC score (clinical scoring system) for subjects with persistent or disseminated primary pulmonary coccidioidomycosis (PPC), Step 2 | Day 180 through Day 365
Quartiles of time to resolution of each symptom contributing to the modified SAnds-PPC score for subjects with primary pulmonary coccidioidomycosis (PPC) from Step 2 | Day 1 through Day 85
Summary statistics for PROMIS Item Bank v2.0 - Ability to Participate in Social Roles and Activities - Short Form 4a for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 1 through Day 365
Summary statistics for the mental component summary (MCS) and the physical component summary (PCS) scores of the SF-12v2 instrument for subjects that are prescribed antifungal therapy vs. no therapy for PPC, Step 2 | Day 1 through Day 365

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Banner - University Medical Center Advanced Lung Disease Clinic - Phoenix, Phoenix, Arizona
  - The University of Arizona - Banner University Medical Center Tucson Campus - Tucson, Tucson, Arizona
  - Kaiser Permanente Chester Avenue Medical Offices - Pulmonology, Bakersfield, California
  - Kern Medical Center, Bakersfield, California
  - UCSF Fresno Center for Medical Education and Research - Clinical Research Center, Fresno, California
  - Kaiser Permanente Antelope Valley Medical Offices - Infectious Diseases, Lancaster, California